CLINICAL TRIAL: NCT05191888
Title: 14-day PCAB-based and Reverse Hybrid Therapy Fro Helicobacter Pylori
Brief Title: 14-day PCAB-based High-dose Dual Therapy and14-day PCAB-based Triple Therapy vs 14-day PPI-based Reverse Hybrid Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, DENG-CHYANG WU, Clinical Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20210136
Record Dates: First submitted 2021-12-28; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Helicobacter Pylori Eradication
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Clarithromycin; Rabeprazole; Metronidazole

STUDY DESIGN:
Intervention Model Description: 1. 14-day vonoprazan high-dose two-in-one therapy
  2. 14-day vonoprazan triple therapy
  3. 14th Rabeprazole reverse mixed therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 14-day vonoprazan high-dose two-in-one therapy (Active Comparator): vonoprazan 20mg bid and amoxicillin 750mg qid
  Interventions: Drug: Vonoprazan and Amoxicillin
- 14-day vonoprazan triple therapy (Active Comparator): vonoprazan 20mg bid and amoxicillin 1gm bid and clarithromycin 500mg bid
  Interventions: Drug: Vonoprazan, Amoxicillin and Clarithromycin
- 14th Rabeprazole reverse mixed therapy (Active Comparator): first 7 days rabeprazole 20mg bid and amoxicillin 1gm bid and clarithromycin 500mg bid and metronidazole 500mg bid Next 7 days rabeprazole 20mg bid and amoxicillin 1gm bid
  Interventions: Drug: Rabeprazole, Amoxicillin, Clarithromycin and Metronidazole

INTERVENTIONS:
Drug: Vonoprazan and Amoxicillin — 14-day vonoprazan high-dose two-in-one therapy
  Arms: 14-day vonoprazan high-dose two-in-one therapy
Drug: Vonoprazan, Amoxicillin and Clarithromycin — 14-day vonoprazan triple therapy
  Arms: 14-day vonoprazan triple therapy
Drug: Rabeprazole, Amoxicillin, Clarithromycin and Metronidazole — 14th Rabeprazole reverse mixed therapy
  Arms: 14th Rabeprazole reverse mixed therapy

SUMMARY:
1. Test for Helicobacter pylori. The test items include urease test, histology, bacterial culture, serology, and urea breath test. At least two positive results can be used to confirm the diagnosis.
2. To ensure that the research results are not artificially distorted, this trial is a randomized study. Random allocation (which means that the subjects will use the "random number table generated by a computer similar to the lottery" to determine the treatment group) accept one of the following schemes (1:1:1).

DETAILED DESCRIPTION:
Helicobacter pylori (H.pylori) infect more than 50% of humans globally. This study were (1) to test whether the efficacies of 14-day PCAB-based high-dose dual therapy and 14-day PPI-based reverse hybrid therapy can achieve a higher eradication rate than 14-day PCAB-based triple therapy in the first-line treatment of H pylori infection, (2) to compare the eradication rates of 14-day PCAB-based and PPI-based bismuth quadruple therapies in the second-line treatment of H pylori infection, and (3) to examine the impacts of antibiotic resistance of H pylori as well as CYP3A4, CYP2C19 and IL-1B -511 genotypes of host on the eradication efficacies of anti-H pylori treatments.

ELIGIBILITY:
Inclusion Criteria:

Subjects infected with Helicobacter pylori.

Exclusion Criteria:

1. Those who have ever received Helicobacter pylori sterilization treatment.
2. Those who are allergic to the drugs used in this research.
3. Those who have had stomach surgery.
4. Those with severe liver cirrhosis or uremia or malignant tumors.
5. Women who are pregnant or breastfeeding.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 906 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the rate of Helicobacter pylori | 6 week after finishing study drugs
  Evaluate eradication outcome by 13C uear breath test

SECONDARY OUTCOMES:
Adverse drug reactions | 2weeks after finishing study drugs
  drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Hsu PI, Chen CL, Shih CA, Chen KY, Tai WC, Chuah SK, Lee CL, Tsay FW, Yang JC, Lei WY, Kuo CH, Shie CB, Lee HC, Yamaoka Y, Graham DY, Wu DC; Taiwan Acid-related Disease and Microbiota (TARD-M) Consortium. Vonoprazan High-Dose Dual, Vonoprazan Triple, and Rabeprazole Reverse Hybrid Therapies for First-Line Treatment of Helicobacter pylori Infection: A Multicenter Randomized Trial. Am J Gastroenterol. 2025 Jun 16. doi: 10.14309/ajg.0000000000003607. Online ahead of print. PMID 40560185